CLINICAL TRIAL: NCT01913392
Title: Prospective, Clinical Study of the Effect of Bariatric Surgery, Laparoscopic Sleeve Gastrectomy, on the Pharmacokinetics of Immunosuppressive Drugs in the Morbidly Obese, Kidney Transplant Candidate
Brief Title: Effect of Laparoscopic Sleeve Gastrectomy in the Morbidly Obese, Kidney Transplant Candidate
Status: Completed | Type: Observational
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Collaborators: Canadian surgical research fund (Unknown); Astellas Pharma Canada, Inc. (Industry)
Responsible Party: Principal Investigator, Gabriel Chan, Md, Transplant and general surgeon, Maisonneuve-Rosemont Hospital
Other Study IDs: 2014-530-13022
Record Dates: First submitted 2013-07-30; First posted 2013-08-01 (Estimated); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Obesity, Morbid; Transplant; Failure, Kidney
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- morbidly obese, chronic renal disease: adult patients (> 18 years) who have stage 4 or 5 chronic renal disease (CrCl < 30 ml/min) who are being considered for possible future kidney transplantation. The study inclusion criteria are an indication for laparoscopic sleeve gastrectomy (BMI > 40 kg/m2, or BMI > 35 with at least one co-morbidity such as hypertension, dyslipidemia or diabetes)
  Interventions: Procedure: laparoscopic sleeve gastrectomy

INTERVENTIONS:
Procedure: laparoscopic sleeve gastrectomy

SUMMARY:
A prospective clinical trial will study the effects of laparoscopic sleeve gastrectomy in the potential renal transplant candidate who is denied acceptance due mainly to the morbid obesity.

DETAILED DESCRIPTION:
The remaining factor in determining the effectiveness of bariatric surgery in the transplant population will be to study the effect on the pharmacokinetics of immunosuppressive medication, height, weight, BMI, abdominal circumference, blood pressure, Hba1c , average daily insulin requirements, lipid profile, TSH, 24h urine creatinine clearance and the SF-36 Quality of life questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* adult (>18 years)
* stage IV and V chronic renal disease (glomerular filtration rate < 30 ml/min,
* body mass index (BMI) of greater than 40 kg/m2 or > 35 with at least one co-morbidity such as hypertension, dyslipidemia or diabetes

Exclusion Criteria:

* medically unfit for surgical intervention
* previous gastric or intestinal surgery
* active gastric disease
* pregnancy or lactation
* known intolerance to tacrolimus or mycophenolic acid
* awaiting potential multi-organ transplantation
* active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: morbidly obese, kidney transplant candidate with stage IV or V chronic renal disease
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2013-07-18 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
changes in the pharmacokinetics of oral immunosuppressive medications due to bariatric surgery, comparing pre-bariatric surgery to 12 months post-operative | pre-bariatric surgery and 1 year after surgery
  Tacrolimus and Mycophenolate AUC 0-24h
degree of weight loss achieved after bariatric surgery in the chronic renal failure patient. | baseline and every 3 months
  weight, BMI and abdominal circumference measures
Evaluate the change in general quality of life score, SF-36 | Baseline and 1 year after bariatric surgery
  comparison of the SF score between Baseline and month 3, Baseline and month 6 and Baseline and month 12

SECONDARY OUTCOMES:
evaluate changes to residual renal function in the pre-dialysis renal transplant candidate | at baseline versus month 12 post-bariatric surgery
  serum creatinine/ urea, sodium, potassium, magnesium, calcium, phosphate and bicarbonate pre surgery and month 12
evaluate the change in the number and dose of medications required to treat co-morbidities including, hypertension, hyperlipidemia and diabetes mellitus | baseline and 12 month post-bariatric surgery
  concommitant medication records at baseline vs month 12
the incidence of complications post-bariatric surgery will be evaluated | 1, 6 and 12 months post-bariatric surgery
  non serious and serious adverse events collection at Baseline, month 6 and month 12

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Chan, MD, Principal Investigator — Maisonneuve-Rosemont Hospital
Locations (1):
- MaisonneuveRH, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Prospective Study of the Changes in Pharmacokinetics of Immunosuppressive Medications after Laparoscopic Sleeve Gastrectomy — http://doi.org/10.1111/ajt.15602

DOCUMENTS (2):
  • Informed Consent Form (2016-05-26): https://cdn.clinicaltrials.gov/large-docs/92/NCT01913392/ICF_000.pdf
  • Study Protocol (2013-04-18): https://cdn.clinicaltrials.gov/large-docs/92/NCT01913392/Prot_001.pdf